CLINICAL TRIAL: NCT05296018
Title: The Effect of Mandala on Coping With Fatigue, Psychological Well-Being and Stress in Patients Treated With Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Sabahattin Zaim University (Other)
Responsible Party: Principal Investigator, Zülfünaz ÖZER, Principal Investigator, Istanbul Sabahattin Zaim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022-01
Record Dates: First submitted 2022-03-16; First posted 2022-03-25 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Hemodialysis
Keywords: Fatigue; Psychological Well-Being; Stress
MeSH Terms: conditions — Fatigue; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This study is an experimental study with pre-test and post-test control groups
Who Masked: Participant
Masking Description: Single (Participant) Mandala and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mandala (Experimental): Mandala coloring page
  Interventions: Other: Mandala coloring page
- Control group (No Intervention): Routine maintenance will be applied

INTERVENTIONS:
Other: Mandala coloring page — Mandala program will be applied three days a week (30 minutes) for 8 weeks.
  Arms: Mandala

SUMMARY:
The aim of this study is to examine the effect of mandala on coping with fatigue, psychological well-being and stress in patients treated with hemodialysis

DETAILED DESCRIPTION:
The Effect of Mandala on Coping with Fatigue, Psychological Well-Being and Stress in Patients Treated with Hemodialysis

ELIGIBILITY:
Inclusion Criteria:

* be over 18
* Ability to communicate adequately
* Absence of psychiatric problems
* Volunteering to participate in the research
* Receiving hemodialysis treatment for at least 6 months

Exclusion Criteria:

* None

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
The fatigue severity scale | 1. week
  The fatigue severity scale is a measurement of fatigue impact on functioning. It is a short, nine-item self-report questionnaire. Its application is very simple and quick.. Read each statement and circle a number from 1 to 7, based on how accurately it reflects your condition. A total score of less than 36 suggests that you may not be suffering from fatigue. A total score of 36 or more suggests that you may need further evaluation by a physician.
The fatigue severity scale | 4. week
  The fatigue severity scale is a measurement of fatigue impact on functioning. It is a short, nine-item self-report questionnaire. Its application is very simple and quick.. Read each statement and circle a number from 1 to 7, based on how accurately it reflects your condition. A total score of less than 36 suggests that you may not be suffering from fatigue. A total score of 36 or more suggests that you may need further evaluation by a physician.
The fatigue severity scale | 8. week
  The fatigue severity scale is a measurement of fatigue impact on functioning. It is a short, nine-item self-report questionnaire. Its application is very simple and quick.. Read each statement and circle a number from 1 to 7, based on how accurately it reflects your condition. A total score of less than 36 suggests that you may not be suffering from fatigue. A total score of 36 or more suggests that you may need further evaluation by a physician.
The psychological well-being scale | 1. week
  The eight-item Psychological Well-Being Scale identifies important elements of human function, from positive relationships to feelings of efficacy to having a meaningful and purposeful life.This is an 8-item selfreported, 7-point Likert-type measurement scale (1=strongly disagree to 7=strongly agree). Higher scores indicated a higher level of psychological well-being.
The psychological well-being scale | 4. week
  The eight-item Psychological Well-Being Scale identifies important elements of human function, from positive relationships to feelings of efficacy to having a meaningful and purposeful life.This is an 8-item selfreported, 7-point Likert-type measurement scale (1=strongly disagree to 7=strongly agree). Higher scores indicated a higher level of psychological well-being.
The psychological well-being scale | 8. week
  The eight-item Psychological Well-Being Scale identifies important elements of human function, from positive relationships to feelings of efficacy to having a meaningful and purposeful life.This is an 8-item selfreported, 7-point Likert-type measurement scale (1=strongly disagree to 7=strongly agree). Higher scores indicated a higher level of psychological well-being.
The Ways of Coping Inventory (WCI) | 1. week
  The Ways of Coping Inventory (WCI) was developed by Folkman and Lazarus (1980) in order to determine the ways by which individuals cope with general or specific stress situations. The scale is a 30-item likert type scale. The answers to the items of the scale are given in four stages, moving from "does not apply or not used" (0) to "used a great deal" Higher scores in "Self-confident", "Optimistic" and "Seeking of social support" (Approach based coping) mean better coping, and higher scores in "Submissive" and "Helpless styles" (Avoidance based coping) mean worse coping.
The Ways of Coping Inventory (WCI) | 4. week
  The Ways of Coping Inventory (WCI) was developed by Folkman and Lazarus (1980) in order to determine the ways by which individuals cope with general or specific stress situations. The scale is a 30-item likert type scale. The answers to the items of the scale are given in four stages, moving from "does not apply or not used" (0) to "used a great deal" Higher scores in "Self-confident", "Optimistic" and "Seeking of social support" (Approach based coping) mean better coping, and higher scores in "Submissive" and "Helpless styles" (Avoidance based coping) mean worse coping.
The Ways of Coping Inventory (WCI) | 8. week
  The Ways of Coping Inventory (WCI) was developed by Folkman and Lazarus (1980) in order to determine the ways by which individuals cope with general or specific stress situations. The scale is a 30-item likert type scale. The answers to the items of the scale are given in four stages, moving from "does not apply or not used" (0) to "used a great deal" Higher scores in "Self-confident", "Optimistic" and "Seeking of social support" (Approach based coping) mean better coping, and higher scores in "Submissive" and "Helpless styles" (Avoidance based coping) mean worse coping.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul Sabahattin Zaim University, Faculty of Health Sciences, Istanbul, Güneydoğu Anadolu Bölgesi
  - Istanbul Sabahattin Zaim University, Faculty of Health Sciences, Istanbul, Küçükçekmece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Choi H, Hahm SC, Jeon YH, Han JW, Kim SY, Woo JM. The Effects of Mindfulness-Based Mandala Coloring, Made in Nature, on Chronic Widespread Musculoskeletal Pain: Randomized Trial. Healthcare (Basel). 2021 May 28;9(6):642. doi: 10.3390/healthcare9060642. PMID 34071674